CLINICAL TRIAL: NCT00270868
Title: Double Guide Wire Placement Compared With Conventional Method in Cases of Difficult Common Bile Duct Cannulation in Endoscopic Retrograde Cholangiopancreatography Procedures. A Controlled Multicentred Randomized Trial.
Brief Title: Efficacy of Double Wire Technique in Difficult Cases of Common Bile Duct Cannulation in ERCP (UDOGUIA-04)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Puerta de Hierro University Hospital (Other)
Collaborators: Carlos III Health Institute (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PI 04/1942
Record Dates: First submitted 2005-12-27; First posted 2005-12-28 (Estimated); Last update posted 2006-10-18 (Estimated); Status verified 2006-10

CONDITIONS: Bile Duct Diseases
Keywords: Double guide wire technique; Difficult selective biliary cannulation; ERCP; Attempts of cannulation; Post-ERCP complications.
MeSH Terms: conditions — Bile Duct Diseases

INTERVENTIONS:
Procedure: Double guide wire technique
Procedure: Standard bile duct cannulation

SUMMARY:
The purpose of this study is to determine if the double guide wire technique is more effective than the conventional method in those cases of difficult selective biliary cannulation in the ERCP procedures.

DETAILED DESCRIPTION:
Complications associated with ERCP have been related with certain characteristics of the procedure. One is the number of attempts of selective biliary cannulation. Our hypothesis is that double guide wire placement could be a useful technique for selective biliary cannulation in those cases of difficult ERCP procedures, reducing the number of cannulation attempts and the complication associated with the procedure.

We are conducting a controlled prospective multicentre randomized study to compare the double guide wire technique with the conventional method in two groups previously randomized after presenting a difficult selective biliary cannulation under the conventional method. The study is carried out in six public Hospitals from Spain. Assignation is concealed to both groups, and the expected study period is 18 months for a number of randomized patients equal or over 262 (statistical power of 90% with an α-error of 0.05, to detect a success rate of 74% in the group undergoing double guide wire technique against a success rate of 60% in the control group). The main outcome variables are successful selective biliary cannulation (primary outcome variable), number of attempts and morbimortality associated in both groups (secondary outcome variables).

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Clinical and/or radiological suspicion of Bile Duct Diseases which require ERCP procedure with intention of selective biliary cannulation
* Patients must be admitted in the participant hospitals of the investigators units
* Written informed consent of the patient, relative or legal tutor

Exclusion Criteria:

* Previous biliary or pancreatic sphincterotomy
* Previous pneumatic dilatation of duodenal papilla
* Presence of biliary-digestive derivation
* Previous diagnosis or suspected pancreas divisum
* Use of any biliary or pancreatic stent in the last 6 months
* Use of any drug aimed to reduce post-ERCP pancreatitis
* Pregnancy or maternal feeding
* Previous inclusion in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1050
Dates: Start 2004-11; Study Completion 2006-11

PRIMARY OUTCOMES:
Percentage of successful selective biliary cannulation

SECONDARY OUTCOMES:
Number of attempts and time of cannulation.
Morbimortality associated in both groups at hospital discharge and 4 weeks after ERCP procedure
Factors associated with successful cannulation for both techniques

CONTACTS AND LOCATIONS:
Overall Officials: Luis E Abreu, MD, Principal Investigator — Puerta de Hierro University Hospital. Madrid Health Service, Spain
Locations (6):
- Spain (6):
  - León Hospital, León, León
  - Alcorcón Hospital Foundation, Alcorcón, Madrid
  - Puerta de Hierro University Hospital, Madrid, Madrid
  - Navarra Hospital, Pamplona, Navarre
  - Central Hospital of Asturias, Oviedo, Principality of Asturias
  - La Fe University Hospital, Valencia, Valencia

REFERENCES:
- [Background] Classen M, Demling L. [Endoscopic sphincterotomy of the papilla of vater and extraction of stones from the choledochal duct (author's transl)]. Dtsch Med Wochenschr. 1974 Mar 15;99(11):496-7. doi: 10.1055/s-0028-1107790. No abstract available. German. PMID 4835515
- [Background] Cotton PB, Chung SC, Davis WZ, Gibson RM, Ransohoff DF, Strasberg SM. Issues in cholecystectomy and management of duct stones. Am J Gastroenterol. 1994 Aug;89(8 Suppl):S169-76. No abstract available. PMID 8048408
- [Background] Ballinger AB, McHugh M, Catnach SM, Alstead EM, Clark ML. Symptom relief and quality of life after stenting for malignant bile duct obstruction. Gut. 1994 Apr;35(4):467-70. doi: 10.1136/gut.35.4.467. PMID 7513672
- [Background] Sherman S, Lehman GA. Endoscopic therapy of pancreatic disease. Gastroenterologist. 1997 Dec;5(4):262-77. PMID 9436003
- [Background] Cotton PB, Lehman G, Vennes J, Geenen JE, Russell RC, Meyers WC, Liguory C, Nickl N. Endoscopic sphincterotomy complications and their management: an attempt at consensus. Gastrointest Endosc. 1991 May-Jun;37(3):383-93. doi: 10.1016/s0016-5107(91)70740-2. PMID 2070995
- [Background] Freeman ML. Adverse outcomes of endoscopic retrograde cholangiopancreatography. Rev Gastroenterol Disord. 2002 Fall;2(4):147-68. PMID 12481167
- [Background] Freeman ML, Nelson DB, Sherman S, Haber GB, Herman ME, Dorsher PJ, Moore JP, Fennerty MB, Ryan ME, Shaw MJ, Lande JD, Pheley AM. Complications of endoscopic biliary sphincterotomy. N Engl J Med. 1996 Sep 26;335(13):909-18. doi: 10.1056/NEJM199609263351301. PMID 8782497
- [Background] Freeman ML, DiSario JA, Nelson DB, Fennerty MB, Lee JG, Bjorkman DJ, Overby CS, Aas J, Ryan ME, Bochna GS, Shaw MJ, Snady HW, Erickson RV, Moore JP, Roel JP. Risk factors for post-ERCP pancreatitis: a prospective, multicenter study. Gastrointest Endosc. 2001 Oct;54(4):425-34. doi: 10.1067/mge.2001.117550. PMID 11577302
- [Background] Loperfido S, Angelini G, Benedetti G, Chilovi F, Costan F, De Berardinis F, De Bernardin M, Ederle A, Fina P, Fratton A. Major early complications from diagnostic and therapeutic ERCP: a prospective multicenter study. Gastrointest Endosc. 1998 Jul;48(1):1-10. doi: 10.1016/s0016-5107(98)70121-x. PMID 9684657
- [Background] Vandervoort J, Soetikno RM, Tham TC, Wong RC, Ferrari AP Jr, Montes H, Roston AD, Slivka A, Lichtenstein DR, Ruymann FW, Van Dam J, Hughes M, Carr-Locke DL. Risk factors for complications after performance of ERCP. Gastrointest Endosc. 2002 Nov;56(5):652-6. doi: 10.1067/mge.2002.129086. PMID 12397271
- [Background] Masci E, Toti G, Mariani A, Curioni S, Lomazzi A, Dinelli M, Minoli G, Crosta C, Comin U, Fertitta A, Prada A, Passoni GR, Testoni PA. Complications of diagnostic and therapeutic ERCP: a prospective multicenter study. Am J Gastroenterol. 2001 Feb;96(2):417-23. doi: 10.1111/j.1572-0241.2001.03594.x. PMID 11232684
- [Background] Masci E, Mariani A, Curioni S, Testoni PA. Risk factors for pancreatitis following endoscopic retrograde cholangiopancreatography: a meta-analysis. Endoscopy. 2003 Oct;35(10):830-4. doi: 10.1055/s-2003-42614. PMID 14551860
- [Background] Friedland S, Soetikno RM, Vandervoort J, Montes H, Tham T, Carr-Locke DL. Bedside scoring system to predict the risk of developing pancreatitis following ERCP. Endoscopy. 2002 Jun;34(6):483-8. doi: 10.1055/s-2002-32004. PMID 12048633
- [Background] Slivka A. A new technique to assist in bile duct cannulation. Gastrointest Endosc. 1996 Nov;44(5):636. doi: 10.1016/s0016-5107(96)70038-x. No abstract available. PMID 8934189
- [Background] Dumonceau JM, Deviere J, Cremer M. A new method of achieving deep cannulation of the common bile duct during endoscopic retrograde cholangiopancreatography. Endoscopy. 1998 Sep;30(7):S80. doi: 10.1055/s-2007-1001379. No abstract available. PMID 9826155
- [Derived] Herreros de Tejada A, Calleja JL, Diaz G, Pertejo V, Espinel J, Cacho G, Jimenez J, Millan I, Garcia F, Abreu L; UDOGUIA-04 Group. Double-guidewire technique for difficult bile duct cannulation: a multicenter randomized, controlled trial. Gastrointest Endosc. 2009 Oct;70(4):700-9. doi: 10.1016/j.gie.2009.03.031. Epub 2009 Jun 27. PMID 19560764